CLINICAL TRIAL: NCT00446030
Title: A Phase II, Open-Label, Multicenter, Pilot Study of the Safety & Efficacy of Two Docetaxel-Based Regimens Plus Bevacizumab for the Adjuvant Treatment of Subjects With Node Positive or High Risk Node Negative Breast Cancer
Brief Title: Pilot Study of the Safety & Efficacy of Two Docetaxel-Based Regimens Plus Bevacizumab for the Adjuvant Treatment of Subjects With Node Positive or High Risk Node Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOCET_L_00713
Record Dates: First submitted 2007-03-08; First posted 2007-03-12 (Estimated); Results first posted 2011-11-04 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Doxorubicin; Carboplatin; Gemcitabine; Cyclophosphamide; Trastuzumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stratum 1: TAC + Bevacizumab (Experimental): Human epidermal growth factor receptor-2 (HER2) negative participants stratified at registration, were administered chemotherapy with docetaxel, doxorubicin and cyclosphosphamide (TAC) + bevacizumab for Cycles 1-6 (every 3 weeks), and followed with maintenance therapy with bevacizumab every 3 weeks for a total of 52 weeks.
  All participants were administered prophylactic recombinant Granulocyte Colony Stimulating Factor (G-CSF) during chemotherapy, based on a dose recommended by the manufacturer. For participants with estrogen receptor (ER) or progesterone receptor (PR) positive tumors, anti-estrogen therapy was recommended. Participants could receive radiation therapy at the discretion of the treating medical and radiation oncologist.
  Interventions: Drug: Docetaxel; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Bevacizumab
- Stratum 2: TCH + Bevacizumab (Experimental): HER2 positive participants stratified at registration, were administered chemotherapy with docetaxel, carboplatin and trastuzumab (TCH) + bevacizumab for Cycles 1-6 (every 3 weeks), and followed with maintenance therapy with bevacizumab and trastuzumab every 3 weeks for a total of 52 weeks.
  All participants were administered prophylactic recombinant Granulocyte Colony Stimulating Factor (G-CSF) during chemotherapy, based on a dose recommended by the manufacturer. For participants with estrogen receptor (ER) or progesterone receptor (PR) positive tumors, anti-estrogen therapy was recommended. Participants could receive radiation therapy at the discretion of the treating medical and radiation oncologist.
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Drug: Trastuzumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m^2 administered IV on Day 1 for Cycles 1-6
  All participants received a prophylactic steroid regimen prior to each dose of docetaxel - Dexamethasone 8 mg orally 12 hours prior to docetaxel, dexamethasone 10 mg IV just prior the docetaxel infusion and 8 mg orally 12 hours after docetaxel administration. If a participant had not taken their oral dexamethasone the evening prior to receiving docetaxel, the dose of the pre-docetaxel infusion of dexamethasone was increased from 10 mg IV to 15 mg IV. A Dexamethasone 8 mg equivalent may have been used (dexamethasone 8 mg = methylprednisolone 40 mg = prednisone 50 mg = prednisolone 50 mg).
  Other Names: Taxotere®
Drug: Doxorubicin — 50 mg/m^2 administered IV on Day 1 for Cycles 1-6
  Arms: Stratum 1: TAC + Bevacizumab
Drug: Carboplatin — 6 mg/mL/min (target area under the curve [AUC] dose) administered IV on Day 1 for Cycles 1-6
  Other Names: Gemzar®
  Arms: Stratum 2: TCH + Bevacizumab
Drug: Cyclophosphamide — 500 mg/m^2 administered IV on Day 1 for Cycles 1-6
  Arms: Stratum 1: TAC + Bevacizumab
Drug: Trastuzumab — A single loading dose of 8 mg/kg administered IV on Day 2 for Cycle 1, and 6 mg/kg administered IV on Day 1 for Cycles 2-6 and for maintenance therapy
  Arms: Stratum 2: TCH + Bevacizumab
Drug: Bevacizumab — 15 mg/kg administered IV on Day 1 for Cycles 1-6, and for maintenance therapy

SUMMARY:
This is a phase II, open-label, multicenter, pilot study of the safety and efficacy of two Docetaxel-based regimens plus bevacizumab for the adjuvant treatment of participants with node positive or high risk node negative breast cancer.

The primary objective of this study was to evaluate the cardiac safety, and the secondary objectives were to evaluate safety and toxicity of participants treated with bevacizumab ± trastuzumab administered with 2 different docetaxel-based combination regimens.

This study was originally designed to also evaluate disease-free survival (DFS) and overall survival (OS); however, based on a protocol amendment, follow-up was shortened from 10 years to 2 years, and the efficacy endpoints of disease free survival and overall survival were deleted from the protocol.

ELIGIBILITY:
Inclusion Criteria:

Participants who met the following criteria were eligible for this study:

1. Woman aged 18 to 70 years, inclusive
2. Had histologically proven breast cancer with the most recent surgery done for breast cancer up to 60 days prior to study registration
3. Had definitive surgical treatment - either mastectomy, or breast conserving surgery with axillary lymph node dissection (or sentinel lymph node biopsy) for operable breast cancer (T1-3, clinical N0-1, and M0)
4. Must have been either "lymph node positive" or "high risk lymph node negative"

   1. Were lymph node positive participants who had at least 1 axillary lymph node involved by breast cancer. (with lymph node metastasis >0.2 mm)
   2. Were high risk lymph node negative participants had no lymph node involvement and at least 1 of the following factors:

      * tumor size >2 cm
      * estrogen receptor (ER) and progesterone receptor (PR) status negative
      * histologic and/or nuclear Grade 2/3
      * age <35 years
5. Were participants with the Human Epidermal growth factor Receptor 2 (HER2/neu) status (positive or negative) known at the time of signing the informed consent
6. Had the estrogen and progesterone receptor status known prior to study registration
7. Had Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
8. Had normal cardiac function, confirmed by left ventricular ejection fraction (LVEF) or shortening fraction (echocardiography [ECHO] or multiple-gated acquisition [MUGA] scan respectively)
9. Had the following hematology criteria confirmed within 2 weeks prior to study registration:

   * Absolute neutrophil count (ANC) >1,500/microL
   * Platelets >100,000/microL
   * Hemoglobin ≥ 9 g/dL
10. Met hepatic function evaluation criteria for bilirubin and AST levels within 2 weeks prior to study registration
11. Had completed staging work-up within 35 days (within 1 year for mammography or breast magnetic resonance imaging (MRI) prior to study registration
12. May have had MammoSite® brachytherapy radiation when performed immediately following surgery and prior to receiving chemotherapy. The balloon catheter must have been removed at least 28 days prior to the start of study treatment
13. May have had bilateral, synchronous breast cancer provided one primary tumor met the staging criteria
14. Women of child bearing potential must have had a negative pregnancy test within 14 days prior to day 1 cycle 1
15. Had consented to using an effective, non-hormonal method of contraception while receiving study treatment and for at least six (6) months following the last dose of bevacizumab, and must have been advised not to breast feed for at least six (6) months following the last dose of bevacizumab.
16. Signed an informed consent prior to beginning any protocol-specific procedures, and had documented expected cooperation during the study treatment and follow-up periods

Exclusion Criteria:

Participants with the following criteria were excluded from this study:

1. Had prior systemic anticancer therapy for invasive breast cancer (immunotherapy,hormonotherapy, chemotherapy)
2. Had prior anthracycline therapy, taxoids, or platinum salts for any malignancy
3. Had prior radiation therapy for breast cancer or any radiotherapy to the chest wall for any other malignancy
4. Was pregnant or lactating
5. Had pre-existing motor or sensory neurotoxicity of a severity >Grade 2 by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 3.0
6. Had cardiac disease or risk for same as follows:

   * Any documented myocardial infarction
   * Angina pectoris that required the use of anti-anginal medication
   * Any history of documented congestive heart failure
   * Grade 3 or Grade 4 cardiac arrhythmia (NCI CTCAE, version 3.0)
   * Clinically significant valvular heart disease
   * Had cardiomegaly
   * Had poorly controlled hypertension, i.e., diastolic greater than 100 mmHg. (Participants who were well controlled on medication were eligible)
   * Were currently receiving medications administered for cardiac arrhythmia, angina or congestive heart failure (e.g., digitalis, beta-blockers, calcium channel-blockers), that alter cardiac conduction, unless the medications were administered for other reasons (e.g., hypertension)
7. Had other serious illness or medical conditions including

   * History of significant neurologic or psychiatric disorders including psychotic disorders, dementia or seizures that prohibited the understanding and giving of informed consent
   * Active uncontrolled infection
   * Active peptic ulcer
   * Unstable diabetes mellitus
   * with symptomatic, intrinsic lung disease resulting in dyspnoea at rest
   * Clinically significant peripheral vascular disease
   * Evidence of bleeding diathesis or coagulopathy
   * Urine protein:creatinine ratio >1.0 at screening
   * History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, inflammatory bowel disease or other gastrointestinal condition increasing the risk of perforation within 6 months of beginning chemotherapy
   * Serious, non-healing wound, ulcer, or bone fracture
   * Known central nervous system (CNS) disease
   * History of stroke or transient ischemic attack (TIA)
   * Known hepatic cirrhosis
8. Had past or current history of neoplasm other than breast carcinoma, except for:

   * Curatively treated non-melanoma skin cancer
   * In situ carcinoma of the cervix
   * Other cancer curatively treated and with no evidence of disease for at least 10 years
   * Ductal carcinoma in-situ (DCIS) of the breast
   * Lobular carcinoma in-situ (LCIS) of the breast
9. Was currently on therapy with any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulators (SERMs), either for osteoporosis or prevention of breast cancer
10. Had chronic treatment with corticosteroids unless initiated >6 months prior to study registration and at low dose (<20 mg methylprednisolone or equivalent)
11. Had concurrent treatment with ovarian hormonal replacement therapy
12. Had concurrent treatment with other experimental drugs
13. Had concurrent treatment with any other anticancer therapy
14. Was male
15. Had known hypersensitivity to Chinese hamster ovary products or other recombinant human or humanized antibodies and/or hypersensitivity to any of the study drugs or their ingredients (e.g., polysorbate 80 in docetaxel)
16. Had minor surgical procedures within 7 days prior to day 1 of study treatment; or major surgical procedures within 28 days prior to day 1 of study treatment or had any anticipated a surgical procedure during the chemotherapy portion of this study
17. Was directly (or was a relative of the study staff) involved in the conduct of the protocol
18. Had a mental condition or psychiatric disorder rendering her unable to understand the nature, scope, and possible consequences of the study
19. Was unlikely to comply with protocol

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2007-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vicki Erickson, MSN, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States

REFERENCES:
- [Derived] Hurvitz SA, Bosserman LD, Chan D, Hagenstad CT, Kass FC, Smith FP, Rodriguez GI, Childs BH, Slamon DJ. Cardiac safety results from a phase II, open-label, multicenter, pilot study of two docetaxel-based regimens plus bevacizumab for the adjuvant treatment of subjects with node-positive or high-risk node-negative breast cancer. Springerplus. 2014 May 12;3:244. doi: 10.1186/2193-1801-3-244. eCollection 2014. PMID 24860718

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 127 participants were registered for this study, and stratified for treatment based on their HER2 status. 93 participants were in Stratum 1 (HER2 negative) and 34 were in Stratum 2 (HER2 positive). One participant in Stratum 1 discontinued at her own request prior to receiving any treatment, but was allowed to enter follow-up.
Groups:
- Stratum 1: TAC + Bevacizumab: HER2 negative participants were administered chemotherapy with docetaxel, doxorubicin and cyclosphosphamide (TAC) + bevacizumab every 3 weeks for 6 cycles, and maintenance therapy with bevacizumab every 3 weeks for a total of 52 weeks.
- Stratum 2: TCH + Bevacizumab: HER2 positive participants were administered chemotherapy with docetaxel, carboplatin and trastuzumab (TCH) + bevacizumab every 3 weeks for 6 cycles, and maintenance therapy with bevacizumab and trastuzumab every 3 weeks for a total of 52 weeks.
Period: TREATMENT (up to 52 Weeks)
Arm/Group | Stratum 1: TAC + Bevacizumab | Stratum 2: TCH + Bevacizumab
Started | 93 | 34
RECEIVED TREATMENT | 92 | 34
Completed | 49 (Participants who completed treatment) | 25 (Participants who completed treatment)
Not Completed | 44 | 9
Not completed — Adverse Event | 29 | 8
Not completed — Subject Request | 9 | 1
Not completed — Poor compliance | 1 | 0
Not completed — Suspicious meningioma | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Patient concern | 1 | 0
Not completed — No treatment, but went to follow-up | 1 | 0
Period: FOLLOW-UP (up to 2-years)
Arm/Group | Stratum 1: TAC + Bevacizumab | Stratum 2: TCH + Bevacizumab
Started | 93 (All participants, including those who discontinued treatment, continued to the follow-up period.) | 34
Completed | 63 | 25
Not Completed | 30 | 9
Not completed — Subject's request | 9 | 4
Not completed — Poor compliance to protocol | 5 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Death | 2 | 2
Not completed — Disease/Breast cancer recurrence/relapse | 3 | 2
Not completed — Investigator decision to close the study | 2 | 0
Not completed — Per physician discretion | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Patient concern | 1 | 0
Not completed — Right axilla wound | 1 | 0
Not completed — Missed last visit due to hysterectomy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1: TAC + Bevacizumab | Stratum 2: TCH + Bevacizumab | Total
Number analyzed (Participants) | 92 | 34 | 126
Age Continuous [Mean (Standard Deviation); unit: years] | 50.7 (10.9) | 49.9 (9.38) | 50.5 (9.88)
Age, Customized [Number; unit: participants]
  < 65 years | 84 | 33 | 117
  >=65 years | 8 | 1 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 34 | 126
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 82 | 23 | 105
  Black | 2 | 3 | 5
  Asian, Oriental | 2 | 6 | 8
  Unknown or Not Reported | 6 | 2 | 8
weight [Mean (Standard Deviation); unit: kg] | 76.37 (17.590) | 72.09 (14.766) | 75.21 (16.925)
Eastern Cooperative Oncology Group (ECOG) performance status score [Number; unit: Participants] — The ECOG performance status score is used to assess how a patient's disease is progressing and to assess how the disease affects the patient's daily living abilities. The ECOG score ranges from 0-5, with 0 indicating the best outcome and a score of 5 indicating the worst outcome. An ECOG score "0" reflects a fully active patient, able to carry on all pre-disease performance without restriction. An ECOG score "1" reflects a participant restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  Participants
    ECOG Performance Score is 0 | 86 | 30 | 116
    ECOG Performance Score is 1 | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Grade 3/4 Clinical Congestive Heart Failure (CHF)
Description: The percentage of participants with Grade 3/4 clinical CHF was calculated. Grade 3/4 CHF symptoms included cardiac failure congestive, cardiomyopathy, and left ventricular dysfunction (LVEF). Echocardiography (ECG) or multiple-gated acquisition (MUGA) scans were scheduled after Cycles 3 and 6 of chemotherapy, after every 3rd cycle of trastuzumab alone, at end of therapy and every 6 months at follow-up to measure changes in LVEF. Clinical symptoms e.g., shortness of breath, tachycardia, cough, neck vein distention, cardiomegaly, hepatomegaly were further investigated for CHF.
Time Frame: up to 2 years
Population: Safety population - all participants who received at least 1 dose of any study treatment.
Measure: Mean (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Stratum 1: TAC + Bevacizumab | Stratum 2: TCH + Bevacizumab
Number analyzed (Participants) | 92 | 34
Percentage of Participants | 4.3 [1.2 to 10.8] | 0 [0.0 to 10.3]

2. Secondary Outcome: Disease-free Survival (DFS) & Overall Survival (OS) of Participants
Description: DFS is the time from study registration until recurrence of tumor or death from any cause in the absence of previous documentation of tumor recurrence. For participants who are removed from the study follow-up prior to documentation of the tumor recurrence, DFS will be censored at the last date the participant was known to be disease-free.
  OS is the time from date of registration to date of death. In the absence of confirmation of death, survival time will be censored at the last date the participant is known to be alive.
Time Frame: up to 10 years
Population: Based on a protocol amendment
  * this study was shortened from 10 years to 2 years
  * the efficacy endpoints of disease free survival, and overall survival were deleted from the protocol.
  Therefore, no analysis was performed for DFS or OS.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stratum 1: TAC + Bevacizumab | Stratum 2: TCH + Bevacizumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: In the table below for 'other adverse events', the number of participants affected are participants who exhibited one or more of any adverse event.
Arm/Group | Stratum 1: TAC + Bevacizumab | Stratum 2: TCH + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 27/92 | 7/34
Other Adverse Events (participants affected / at risk) | 92/92 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1: TAC + Bevacizumab (N=92) | Stratum 2: TCH + Bevacizumab (N=34)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 4 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 2
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
DUODENAL ULCER (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0
NEUTROPENIC COLITIS (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0
ADVERSE DRUG REACTION (General disorders) | 1 | 0
IMPAIRED HEALING (General disorders) | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 2 | 0
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 | 0
NEUTROPENIC INFECTION (Infections and infestations) | 1 | 0
PERIRECTAL ABSCESS (Infections and infestations) | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 0 | 1
NEUTROPENIC SEPSIS (Infections and infestations) | 0 | 1
PERIDIVERTICULAR ABSCESS (Infections and infestations) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 0
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 1 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 1
HYDROCEPHALUS (Nervous system disorders) | 0 | 1
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 0 | 1
MOOD ALTERED (Psychiatric disorders) | 0 | 1
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1: TAC + Bevacizumab (N=92) | Stratum 2: TCH + Bevacizumab (N=34)
NEUTROPENIA (Blood and lymphatic system disorders) | 36 | 5
ANAEMIA (Blood and lymphatic system disorders) | 33 | 13
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 25 | 11
LEUKOPENIA (Blood and lymphatic system disorders) | 19 | 5
LYMPHOPENIA (Blood and lymphatic system disorders) | 6 | 1
TACHYCARDIA (Cardiac disorders) | 11 | 3
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 5 | 1
EAR PAIN (Ear and labyrinth disorders) | 5 | 0
HEARING IMPAIRED (Ear and labyrinth disorders) | 1 | 2
TINNITUS (Ear and labyrinth disorders) | 1 | 2
LACRIMATION INCREASED (Eye disorders) | 31 | 14
DRY EYE (Eye disorders) | 11 | 3
VISION BLURRED (Eye disorders) | 11 | 5
NAUSEA (Gastrointestinal disorders) | 75 | 28
DIARRHOEA (Gastrointestinal disorders) | 57 | 24
CONSTIPATION (Gastrointestinal disorders) | 46 | 18
VOMITING (Gastrointestinal disorders) | 39 | 12
STOMATITIS (Gastrointestinal disorders) | 30 | 12
DYSPEPSIA (Gastrointestinal disorders) | 24 | 13
ABDOMINAL PAIN (Gastrointestinal disorders) | 16 | 4
HAEMORRHOIDS (Gastrointestinal disorders) | 10 | 3
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 9 | 4
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 7 | 2
DRY MOUTH (Gastrointestinal disorders) | 6 | 3
GINGIVAL BLEEDING (Gastrointestinal disorders) | 6 | 2
ORAL PAIN (Gastrointestinal disorders) | 6 | 2
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 5 | 2
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 5 | 2
GASTRITIS (Gastrointestinal disorders) | 0 | 2
FATIGUE (General disorders) | 79 | 30
MUCOSAL INFLAMMATION (General disorders) | 16 | 7
ASTHENIA (General disorders) | 15 | 4
PYREXIA (General disorders) | 15 | 3
PAIN (General disorders) | 14 | 5
OEDEMA PERIPHERAL (General disorders) | 11 | 7
CHEST DISCOMFORT (General disorders) | 7 | 2
CHEST PAIN (General disorders) | 5 | 1
CHILLS (General disorders) | 3 | 3
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 3
FEELING HOT (General disorders) | 0 | 2
DRUG HYPERSENSITIVITY (Immune system disorders) | 2 | 2
HYPERSENSITIVITY (Immune system disorders) | 0 | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 13 | 5
NASOPHARYNGITIS (Infections and infestations) | 12 | 1
RHINITIS (Infections and infestations) | 12 | 4
SINUSITIS (Infections and infestations) | 11 | 7
URINARY TRACT INFECTION (Infections and infestations) | 10 | 8
CANDIDIASIS (Infections and infestations) | 5 | 1
HERPES ZOSTER (Infections and infestations) | 5 | 1
LARYNGITIS (Infections and infestations) | 5 | 3
ORAL CANDIDIASIS (Infections and infestations) | 4 | 2
CATHETER SITE INFECTION (Infections and infestations) | 1 | 2
FOLLICULITIS (Infections and infestations) | 1 | 3
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 10 | 4
CONTUSION (Injury, poisoning and procedural complications) | 4 | 3
WEIGHT DECREASED (Investigations) | 10 | 4
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 | 6
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 4 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 7
EJECTION FRACTION DECREASED (Investigations) | 3 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 38 | 10
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 13 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 12 | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 47 | 20
BONE PAIN (Musculoskeletal and connective tissue disorders) | 31 | 5
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 20 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 18 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 14 | 7
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 13 | 8
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 10 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 6 | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 | 5
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 2 | 2
HEADACHE (Nervous system disorders) | 40 | 16
DYSGEUSIA (Nervous system disorders) | 25 | 17
NEUROPATHY PERIPHERAL (Nervous system disorders) | 18 | 4
DIZZINESS (Nervous system disorders) | 11 | 4
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 8 | 5
MEMORY IMPAIRMENT (Nervous system disorders) | 5 | 2
PARAESTHESIA (Nervous system disorders) | 5 | 3
SYNCOPE (Nervous system disorders) | 4 | 2
AMNESIA (Nervous system disorders) | 2 | 2
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 0 | 2
HYPERAESTHESIA (Nervous system disorders) | 0 | 2
INSOMNIA (Psychiatric disorders) | 39 | 16
DEPRESSION (Psychiatric disorders) | 19 | 6
ANXIETY (Psychiatric disorders) | 18 | 5
CONFUSIONAL STATE (Psychiatric disorders) | 2 | 3
DYSURIA (Renal and urinary disorders) | 5 | 3
PROTEINURIA (Renal and urinary disorders) | 5 | 3
HAEMATURIA (Renal and urinary disorders) | 2 | 3
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 7 | 4
AMENORRHOEA (Reproductive system and breast disorders) | 5 | 2
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 4 | 2
BREAST DISCOMFORT (Reproductive system and breast disorders) | 1 | 2
BREAST PAIN (Reproductive system and breast disorders) | 1 | 2
BREAST TENDERNESS (Reproductive system and breast disorders) | 1 | 2
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 3
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 43 | 18
COUGH (Respiratory, thoracic and mediastinal disorders) | 30 | 8
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 22 | 7
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 17 | 10
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 15 | 3
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 7 | 1
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 6 | 6
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 4 | 3
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2 | 2
ALOPECIA (Skin and subcutaneous tissue disorders) | 73 | 28
ERYTHEMA (Skin and subcutaneous tissue disorders) | 14 | 3
RASH (Skin and subcutaneous tissue disorders) | 14 | 9
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 9 | 8
DRY SKIN (Skin and subcutaneous tissue disorders) | 8 | 8
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 6 | 4
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 5 | 3
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 6
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 3 | 2
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 2 | 2
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 | 2
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 | 2
HOT FLUSH (Vascular disorders) | 33 | 15
HYPERTENSION (Vascular disorders) | 26 | 11
LYMPHOEDEMA (Vascular disorders) | 5 | 2
FLUSHING (Vascular disorders) | 3 | 2

LIMITATIONS AND CAVEATS:
The number of participants enrolled into the TCH with bevacizumab arm was reduced to half of the originally intended number. Therefore, all conclusions related to the safety of TCH with bevacizumab must be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to independently publish study results from his site after a multicenter publication, or 12 months after the completion of the study by all sites. He must provide the sponsor a copy of any such publication derived from the study for review and comment at least 60 days in advance of any submission for publication. The Sponsor may request for the publication to be delayed for a limited time, not to exceed 90 days to preserve its proprietary rights.